CLINICAL TRIAL: NCT03930160
Title: Logistic Organ Dysfunction System Role in Predicting 30-day Mortality Outcome in Intensive Care Unit of dr. Cipto Mangunkusumo General Hospital Patients
Brief Title: LODS Role in Predicting 30-day Mortality Outcome in ICU
Status: Completed | Type: Observational
Sponsor: Indonesia University (Other)
Responsible Party: Principal Investigator, Dita Aditianingsih, MD, PhD, Anesthesiologist Consultant, Indonesia University
Other Study IDs: IndonesiaUAnes035
Record Dates: First submitted 2019-04-24; First posted 2019-04-29 (Actual); Last update posted 2019-04-29 (Actual); Status verified 2019-04

CONDITIONS: Mortality
Keywords: Intensive care unit; Logistic Organ Dysfunction System; 30-day Mortality; Sepsis; Mortality prediction
MeSH Terms: conditions — Sepsis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Mortality outcome
  Interventions: Other: Logistic Organ Dysfunction System Score

INTERVENTIONS:
Other: Logistic Organ Dysfunction System Score — Variables of logistic organ dysfunction system score, including: GCS; heart rate; systolic BP; blood urea; serum creatinine; urine output; leucocyte count; platelet count; PaO2/FiO2; serum bilirubin; prothrombin time.
  Other Names: LODS

SUMMARY:
LODS score for deceased ICU patients within 30 days is higher than survived ICU patients

ELIGIBILITY:
Inclusion Criteria:

* adult patient (age 18 years and above) admitted to ICU

Exclusion Criteria:

* patients admitted to ICU due to burn injury, coronary artery disease, post cardiac surgery
* patients with incomplete required information for LODS score
* patients deceased or discharged less than 24 hours of admission

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: intensive care unit patients medical records
Sampling Method: Non-Probability Sample
Enrollment: 439 (Actual)
Dates: Start 2018-05-17 (Actual); Primary Completion 2018-08-17 (Actual); Study Completion 2018-11-23 (Actual)

PRIMARY OUTCOMES:
LODS score discrimination ability | 30 days from admission
  LODS score ability to discriminate patient outcomes based on variables of logistic organ dysfunction system scores: GCS; heart rate; systolic BP; blood urea; serum creatinine; urine output; leucocyte count; platelet count; PaO2/FiO2; serum bilirubin; prothrombin time.
LODS score calibration | 30 days from admission
  LODS score ability to predict patient outcomes based on variables of logistic organ dysfunction system scores: GCS; heart rate; systolic BP; blood urea; serum creatinine; urine output; leucocyte count; platelet count; PaO2/FiO2; serum bilirubin; prothrombin time.
Correlation between LODS score variables with patient outcome | 30 days from admission
  Correlation between patient outcomes with each LODS score variables: GCS; heart rate; systolic BP; blood urea; serum creatinine; urine output; leucocyte count; platelet count; PaO2/FiO2; serum bilirubin; prothrombin time.

SECONDARY OUTCOMES:
Patient outcome | 30 days from admission
  Patient outcome within 30 days of admission to intensive care unit (ICU): deceased or survived
LODS neurologic variable score: Glasgow Coma Scale (GCS) | Day 1
  The score for GCS variable cutoff:
  0 point for 14-15;
  1 point for 9-13; 3 points for 6-8; 5 points for 3-5.
LODS cardiovascular variable score: Heart rate (HR) and/or systolic blood pressure (SBP) | Day 1
  The score for HR (in bpm) and/or SBP (in mmHg) variable cutoff:
  0 point for HR 30-139 and SBP 90-239;
  1 point for SBP 70-89 or 240-269 or HR >=140; 3 points for SBP 40-69 or >=270; 5 points for HR <30 or SBP <40.
LODS renal variable score: serum urea nitrogen (BUN) and/or creatinine and/or urine output (UO) | Day 1
  The score for BUN (in mg/dL) and/or creatinine (in mg/dL) and/or UO (in litres/day) variable cutoff:
  0 point for BUN <17 AND creatinine <1.20 AND UO 0.75-9.99;
  1 point for BUN 17-<28 OR creatinine 1.20-1.59; 3 points for BUN 28-<56 AND creatinine <1.60 AND UO 0.5-0.74 or >=10; 5 points for BUN >=56 OR UO 0.5.
LODS pulmonary variable score: Partial oxygen pressure (PaO2)/Fraction of inspired oxygen (FiO2) on Mechanical Ventilation (MV) or Continuous Positive Airway Pressure (CPAP) | Day 1
  The score for PaO2/FiO2 (in mmHg/%) variable cutoff:
  0 point for no ventilation and no CPAP;
  1 point for >=150; 3 points for <150.
LODS hematologic variable score: white blood cell (WBC) count and/or platelet count | Day 1
  The score for WBC (in x10^3/L) and/or platelet count in (x10^3/L) variable cutoff:
  0 point for WBC 2.5-49.9 and platelet >=50;
  1 point for WBC 1.0-2.4 or >=50.0 OR platelet <50; 3 points for WBC <1.0
LODS hepatic function variable score: Serum Bilirubin and/or Prothrombin time (PT) | Day 1
  The score for serum bilirubin (in mg/dL) and/or PT (in % of standard) variable cutoff:
  0 point for bilirubin <2.0 and PT >=25;
  1 point for bilirubin >=2.0 OR PT<25% or >3.

CONTACTS AND LOCATIONS:
Locations (1):
- Rumah Sakit Cipto Mangunkusumo, Jakarta Pusat, DKI Jakarta, Indonesia

REFERENCES:
- [Background] Power GS, Harrison DA. Why try to predict ICU outcomes? Curr Opin Crit Care. 2014 Oct;20(5):544-9. doi: 10.1097/MCC.0000000000000136. PMID 25159474
- [Background] Rapsang AG, Shyam DC. Scoring systems in the intensive care unit: A compendium. Indian J Crit Care Med. 2014 Apr;18(4):220-8. doi: 10.4103/0972-5229.130573. PMID 24872651
- [Background] Purnama Dewi O, Nurfitri E. Pediatric logistic organ dysfunction score as a predictive tool of dengue shock syndrome outcomes. Paediatrica Indonesiana. 2012;52(2):72-77.
- [Background] Grenvik A, Ayres SM, Holbrook PR, Shoemaker WC, editors. Textbook of Critical Care. Subsequent edition. Philadelphia: W B Saunders Co; 2000. 2227 p
- [Background] Rao SM, Suhasini T. Organization of intensive care unit and predicting outcome of critical illness. Indian J Anaesth. 2003;47(5):328-37.
- [Background] Le Gall JR, Klar J, Lemeshow S, Saulnier F, Alberti C, Artigas A, Teres D. The Logistic Organ Dysfunction system. A new way to assess organ dysfunction in the intensive care unit. ICU Scoring Group. JAMA. 1996 Sep 11;276(10):802-10. doi: 10.1001/jama.276.10.802. PMID 8769590
- [Background] Heldwein MB, Badreldin AM, Doerr F, Lehmann T, Bayer O, Doenst T, Hekmat K. Logistic Organ Dysfunction Score (LODS): a reliable postoperative risk management score also in cardiac surgical patients? J Cardiothorac Surg. 2011 Sep 16;6:110. doi: 10.1186/1749-8090-6-110. PMID 21923900
- [Background] Kim TK, Yoon JR. Comparison of the predictive power of the LODS and APACHE II scoring systems in a neurological intensive care unit. J Int Med Res. 2012;40(2):777-86. doi: 10.1177/147323001204000244. PMID 22613443
- [Background] Saranya AVR S. Comparison of Different Scoring Systems Used in the Intensive Care Unit. Journal of Pulmonary & Respiratory Medicine. 2015;05(04).
- [Background] Timsit JF, Fosse JP, Troche G, De Lassence A, Alberti C, Garrouste-Orgeas M, Azoulay E, Chevret S, Moine P, Cohen Y. Accuracy of a composite score using daily SAPS II and LOD scores for predicting hospital mortality in ICU patients hospitalized for more than 72 h. Intensive Care Med. 2001 Jun;27(6):1012-21. doi: 10.1007/s001340100961. PMID 11497133
- [Background] Timsit JF, Fosse JP, Troche G, De Lassence A, Alberti C, Garrouste-Orgeas M, Bornstain C, Adrie C, Cheval C, Chevret S; OUTCOMEREA Study Group, France. Calibration and discrimination by daily Logistic Organ Dysfunction scoring comparatively with daily Sequential Organ Failure Assessment scoring for predicting hospital mortality in critically ill patients. Crit Care Med. 2002 Sep;30(9):2003-13. doi: 10.1097/00003246-200209000-00009. PMID 12352033
- [Background] Bouch DC, Thompson JP. Severity scoring systems in the critically ill. Contin Educ Anaesth Crit Care Pain. 2008;8:181-5.
- [Background] Dolejs J, Maresova P. Onset of mortality increase with age and age trajectories of mortality from all diseases in the four Nordic countries. Clin Interv Aging. 2017 Jan 21;12:161-173. doi: 10.2147/CIA.S119327. eCollection 2017. PMID 28176929
- [Background] Ingraham AM, Cohen ME, Raval MV, Ko CY, Nathens AB. Comparison of hospital performance in emergency versus elective general surgery operations at 198 hospitals. J Am Coll Surg. 2011 Jan;212(1):20-28.e1. doi: 10.1016/j.jamcollsurg.2010.09.026. PMID 21184955
- [Background] Ball IM, Bagshaw SM, Burns KE, Cook DJ, Day AG, Dodek PM, Kutsogiannis DJ, Mehta S, Muscedere JG, Turgeon AF, Stelfox HT, Wells GA, Stiell IG. Outcomes of elderly critically ill medical and surgical patients: a multicentre cohort study. Can J Anaesth. 2017 Mar;64(3):260-269. doi: 10.1007/s12630-016-0798-4. Epub 2016 Dec 27. PMID 28028673
- [Background] De Jong A, Verzilli D, Sebbane M, Monnin M, Belafia F, Cisse M, Conseil M, Carr J, Jung B, Chanques G, Molinari N, Jaber S. Medical Versus Surgical ICU Obese Patient Outcome: A Propensity-Matched Analysis to Resolve Clinical Trial Controversies. Crit Care Med. 2018 Apr;46(4):e294-e301. doi: 10.1097/CCM.0000000000002954. PMID 29293153
- [Background] Arihan O, Wernly B, Lichtenauer M, Franz M, Kabisch B, Muessig J, Masyuk M, Lauten A, Schulze PC, Hoppe UC, Kelm M, Jung C. Blood Urea Nitrogen (BUN) is independently associated with mortality in critically ill patients admitted to ICU. PLoS One. 2018 Jan 25;13(1):e0191697. doi: 10.1371/journal.pone.0191697. eCollection 2018. PMID 29370259
- [Background] Hashemian SM, Jamaati H, Farzanegan Bidgoli B, Farrokhi FR, Malekmohammad M, Roozdar S, Mohajerani SA, Bagheri A, Radmnand G, Hatami B, Chitsazan M. Outcome of Acute Kidney Injury in Critical Care Unit, Based on AKI Network. Tanaffos. 2016;15(2):89-95. PMID 27904540
- [Background] Engoren M, Maile MD, Heung M, Jewell ES, Vahabzadeh C, Haft JW, Kheterpal S. The Association Between Urine Output, Creatinine Elevation, and Death. Ann Thorac Surg. 2017 Apr;103(4):1229-1237. doi: 10.1016/j.athoracsur.2016.07.036. Epub 2016 Oct 4. PMID 27717425
- [Background] Macedo E, Malhotra R, Bouchard J, Wynn SK, Mehta RL. Oliguria is an early predictor of higher mortality in critically ill patients. Kidney Int. 2011 Oct;80(7):760-7. doi: 10.1038/ki.2011.150. Epub 2011 Jun 29. PMID 21716258
- [Background] Zhang Z, Xu X, Ni H, Deng H. Urine output on ICU entry is associated with hospital mortality in unselected critically ill patients. J Nephrol. 2014 Feb;27(1):65-71. doi: 10.1007/s40620-013-0024-1. Epub 2014 Jan 15. PMID 24424722
- [Background] Saygitov RT, Glezer MG, Semakina SV. Blood urea nitrogen and creatinine levels at admission for mortality risk assessment in patients with acute coronary syndromes. Emerg Med J. 2010 Feb;27(2):105-9. doi: 10.1136/emj.2008.068155. PMID 20156860
- [Background] Teasdale G, Jennett B. Assessment of coma and impaired consciousness. A practical scale. Lancet. 1974 Jul 13;2(7872):81-4. doi: 10.1016/s0140-6736(74)91639-0. No abstract available. PMID 4136544
- [Background] Ting HW, Chen MS, Hsieh YC, Chan CL. Good mortality prediction by Glasgow Coma Scale for neurosurgical patients. J Chin Med Assoc. 2010 Mar;73(3):139-43. doi: 10.1016/S1726-4901(10)70028-9. PMID 20230998
- [Background] Nik A, Sheikh Andalibi MS, Ehsaei MR, Zarifian A, Ghayoor Karimiani E, Bahadoorkhan G. The Efficacy of Glasgow Coma Scale (GCS) Score and Acute Physiology and Chronic Health Evaluation (APACHE) II for Predicting Hospital Mortality of ICU Patients with Acute Traumatic Brain Injury. Bull Emerg Trauma. 2018 Apr;6(2):141-145. doi: 10.29252/beat-060208. PMID 29719845
- [Background] Zhang D, Shen X, Qi X. Resting heart rate and all-cause and cardiovascular mortality in the general population: a meta-analysis. CMAJ. 2016 Feb 16;188(3):E53-E63. doi: 10.1503/cmaj.150535. Epub 2015 Nov 23. PMID 26598376
- [Background] Reunanen A, Karjalainen J, Ristola P, Heliovaara M, Knekt P, Aromaa A. Heart rate and mortality. J Intern Med. 2000 Feb;247(2):231-9. doi: 10.1046/j.1365-2796.2000.00602.x. PMID 10692086
- [Background] Prasada S, Oswalt C, Yeboah P, Saylor G, Bowden D, Yeboah J. Heart rate is an independent predictor of all-cause mortality in individuals with type 2 diabetes: The diabetes heart study. World J Diabetes. 2018 Jan 15;9(1):33-39. doi: 10.4239/wjd.v9.i1.33. PMID 29359027
- [Background] Tongyoo S, Permpikul C, Haemin R, Epichath N. Predicting factors, incidence and prognosis of cardiac arrhythmia in medical, non-acute coronary syndrome, critically ill patients. J Med Assoc Thai. 2013 Feb;96 Suppl 2:S238-45. PMID 23590048
- [Background] Li C, Chen Y, Zheng Q, Wu W, Chen Z, Song L, An S, Li Z, Chen S, Wu SL. Relationship between systolic blood pressure and all-cause mortality: a prospective study in a cohort of Chinese adults. BMC Public Health. 2018 Jan 5;18(1):107. doi: 10.1186/s12889-017-4965-5. PMID 29304766
- [Background] Lv YB, Gao X, Yin ZX, Chen HS, Luo JS, Brasher MS, Kraus VB, Li TT, Zeng Y, Shi XM. Revisiting the association of blood pressure with mortality in oldest old people in China: community based, longitudinal prospective study. BMJ. 2018 Jun 5;361:k2158. doi: 10.1136/bmj.k2158. PMID 29871897
- [Background] Ruggiero C, Metter EJ, Cherubini A, Maggio M, Sen R, Najjar SS, Windham GB, Ble A, Senin U, Ferrucci L. White blood cell count and mortality in the Baltimore Longitudinal Study of Aging. J Am Coll Cardiol. 2007 May 8;49(18):1841-50. doi: 10.1016/j.jacc.2007.01.076. Epub 2007 Apr 23. PMID 17481443
- [Background] Bonaccio M, Di Castelnuovo A, Costanzo S, De Curtis A, Donati MB, Cerletti C, de Gaetano G, Iacoviello L; MOLI-SANI Investigators. Age-sex-specific ranges of platelet count and all-cause mortality: prospective findings from the MOLI-SANI study. Blood. 2016 Mar 24;127(12):1614-6. doi: 10.1182/blood-2016-01-692814. Epub 2016 Feb 10. No abstract available. PMID 26864338
- [Background] Tsai MT, Chen YT, Lin CH, Huang TP, Tarng DC; Taiwan Geriatric Kidney Disease Research Group. U-shaped mortality curve associated with platelet count among older people: a community-based cohort study. Blood. 2015 Sep 24;126(13):1633-5. doi: 10.1182/blood-2015-06-654764. Epub 2015 Aug 11. No abstract available. PMID 26265696
- [Background] van der Bom JG, Heckbert SR, Lumley T, Holmes CE, Cushman M, Folsom AR, Rosendaal FR, Psaty BM. Platelet count and the risk for thrombosis and death in the elderly. J Thromb Haemost. 2009 Mar;7(3):399-405. doi: 10.1111/j.1538-7836.2008.03267.x. Epub 2008 Dec 20. PMID 19143922
- [Background] Ishizuka M, Tago K, Kubota K. Impact of prothrombin time-International Normalized Ratio on outcome of patients with septic shock receiving polymyxin B cartridge hemoperfusion. Surgery. 2014 Jul;156(1):168-75. doi: 10.1016/j.surg.2014.03.009. Epub 2014 Mar 15. PMID 24929766
- [Background] Benediktsson S, Frigyesi A, Kander T. Routine coagulation tests on ICU admission are associated with mortality in sepsis: an observational study. Acta Anaesthesiol Scand. 2017 Aug;61(7):790-796. doi: 10.1111/aas.12918. PMID 28681428
- [Background] Yokoyama Y, Ebata T, Igami T, Sugawara G, Ando M, Nagino M. Predictive power of prothrombin time and serum total bilirubin for postoperative mortality after major hepatectomy with extrahepatic bile duct resection. Surgery. 2014 Mar;155(3):504-11. doi: 10.1016/j.surg.2013.08.022. Epub 2013 Nov 25. PMID 24287146
- [Background] Pierrakos C, Velissaris D, Felleiter P, Antonelli M, Vanhems P, Sakr Y, Vincent JL; EPIC II investigators. Increased mortality in critically ill patients with mild or moderate hyperbilirubinemia. J Crit Care. 2017 Aug;40:31-35. doi: 10.1016/j.jcrc.2017.01.017. Epub 2017 Feb 13. PMID 28314169
- [Background] Su HH, Kao CM, Lin YC, Lin YC, Kao CC, Chen HH, Hsu CC, Chen KC, Peng CC, Wu MS. Relationship between serum total bilirubin levels and mortality in uremia patients undergoing long-term hemodialysis: A nationwide cohort study. Atherosclerosis. 2017 Oct;265:155-161. doi: 10.1016/j.atherosclerosis.2017.09.001. Epub 2017 Sep 4. PMID 28892712
- [Background] Yang TL, Lin YC, Lin YC, Huang CY, Chen HH, Wu MS. Total Bilirubin in Prognosis for Mortality in End-Stage Renal Disease Patients on Peritoneal Dialysis Therapy. J Am Heart Assoc. 2017 Dec 23;6(12):e007507. doi: 10.1161/JAHA.117.007507. PMID 29275374
- [Background] Esteve F, Lopez-Delgado JC, Javierre C, Skaltsa K, Carrio ML, Rodriguez-Castro D, Torrado H, Farrero E, Diaz-Prieto A, Ventura JL, Manez R. Evaluation of the PaO2/FiO2 ratio after cardiac surgery as a predictor of outcome during hospital stay. BMC Anesthesiol. 2014 Sep 26;14:83. doi: 10.1186/1471-2253-14-83. PMID 25928646
- [Background] Villar J, Blanco J, del Campo R, Andaluz-Ojeda D, Diaz-Dominguez FJ, Muriel A, Corcoles V, Suarez-Sipmann F, Tarancon C, Gonzalez-Higueras E, Lopez J, Blanch L, Perez-Mendez L, Fernandez RL, Kacmarek RM; Spanish Initiative for Epidemiology, Stratification & Therapies for ARDS (SIESTA) Network. Assessment of PaO(2)/FiO(2) for stratification of patients with moderate and severe acute respiratory distress syndrome. BMJ Open. 2015 Mar 27;5(3):e006812. doi: 10.1136/bmjopen-2014-006812. PMID 25818272
- [Background] Fialkow L, Farenzena M, Wawrzeniak IC, Brauner JS, Vieira SR, Vigo A, Bozzetti MC. Mechanical ventilation in patients in the intensive care unit of a general university hospital in southern Brazil: an epidemiological study. Clinics (Sao Paulo). 2016 Mar;71(3):144-51. doi: 10.6061/clinics/2016(03)05. PMID 27074175